CLINICAL TRIAL: NCT02157935
Title: A Phase IIIB, 6-Month, Double-blind, Double-dummy, Randomized, Parallel-group, Multicenter Exacerbation Study of Symbicort® Pressurized Metered-Dose Inhaler (pMDI) 160/4.5 μg x 2 Actuations Twice-daily Compared to Formoterol Turbuhaler 4.5 μg x 2 Inhalations Twice-daily in Cronic Obstructive Pulmonary Disease (COPD) Patients.
Brief Title: Comparing the Efficacy of Symbicort® pMDI and Formoterol Turbuhaler in Reducing Exacerbations in Patients With Cronic Obstructive Pulmonary Disease
Acronym: RISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D589UC00001
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: COPD Patients
Keywords: COPD, turbuhaler, pMDI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort pMDI (Active Comparator): Symbicort pMDI, budesonide/formoterol, 160/4.5 μg x 2 actuations BID, for oral inhalation
  Interventions: Drug: Symbicort; Other: Placebo for Symbicort pMDI
- Formoterol Turbuhaler (Active Comparator): Formoterol Turbuhaler, 4.5 μg x 2 actuations BID, for oral inhalation
  Interventions: Drug: Formoterol turbohaler; Other: Placebo for Formoterol Turbohaler

INTERVENTIONS:
Drug: Symbicort — Budesonide/formoterol pMDI, 160/4.5 μg x 2 actuations BID, for oral inhalation, 120 doses
  Arms: Symbicort pMDI
Drug: Formoterol turbohaler — Formoterol Turbuhaler 4.5 μg x 2 actuations BID, for oral inhalation, 60 doses
  Arms: Formoterol Turbuhaler
Other: Placebo for Symbicort pMDI — pMDI, aerosol for oral inhalation, placebo, 120 doses
  Arms: Symbicort pMDI
Other: Placebo for Formoterol Turbohaler — PLacebo powder for oral inhalation, 60 doses
  Arms: Formoterol Turbuhaler

SUMMARY:
Comparing the efficacy of Symbicort® pMDI and Formoterol Turbuhaler in reducing exacerbations in patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
A Phase IIIB, 6-Month, Double-blind, Double-dummy, Randomized, Parallel-group, Multicenter Exacerbation Study of Symbicort® pMDI 160/4.5 μg x 2 Actuations Twice-daily Compared to Formoterol Turbuhaler 4.5 μg x 2 Inhalations Twice-daily in COPD Patients.

ELIGIBILITY:
Inclusion Criteria:

3. A current clinical diagnosis of COPD with COPD symptoms for more than 1 year, according to the GOLD guidelines.

4. Current or previous smoker with a smoking history equivalent to 10 or more pack years (1 pack year = 20 cigarettes smoked per day for 1 year).

5. Post-bronchodilator FEV1/forced vital capacity (FVC) <0.7 (70%) and FEV1 ≤70% of predicted normal (PN) value.

6. Documented use of a short-acting inhaled bronchodilator (β2-agonists or anticholinergics) as rescue medication within 6 months prior to study start.

7. A score of ≥2 on the modified medical research council (MMRC) dyspnea scale. 8. Documented history of ≥1 moderate or severe COPD exacerbation(s) that required treatment with systemic (oral, IM, IV) corticosteroids (a minimum 3 day course of an oral corticosteroid treatment or single depot corticosteroid injection), or hospitalization (defined as an inpatient stay or >24 hour stay in an observation area in the emergency department or other equivalent facility depending on the country and healthcare system) within 2-52 weeks before Visit 1 (i.e., not within the 14 days prior to Visit 1). A history of an exacerbation treated exclusively with antibiotics will not be considered adequate.

Exclusion Criteria:

1. A history of asthma at or after 18 years of age.
2. Subjects with significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure (including significant cor pulmonale), uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator.
3. Known homozygous alpha-1 antitrypsin deficiency.
4. Any significant disease or disorder (e.g., gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study.
5. A history of malignancy (except basal cell carcinoma) within the past 5 years.
6. Active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung disease, or other active pulmonary diseases.
7. Subjects who have needed additions or alterations to their usual maintenance or change in formulation of rescue therapy for COPD due to worsening symptoms within the 14 days prior to Visit 1 and up to Visit 3.
8. CXR (frontal and lateral) with suspicion of pneumonia or other condition/abnormality that will require additional investigation/treatment, or put the subject at risk because of participation in the study.
9. Risk factors for pneumonia: immune suppression (HIV, lupus) or other risk for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's disease, myasthenia gravis, etc.).
10. Pneumonia not resolved within 14 days of Visit 1.
11. Moderate or severe COPD exacerbation that has not resolved within 14 days prior to Visit 1 or a moderate or severe COPD exacerbation that occurs between Visit 1 and Visit 2.
12. Long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day.
13. Subjects who are currently in the intensive rehabilitation phase or scheduled to begin new participation (intensive rehabilitation phase) in a pulmonary rehabilitation program during the study or have started a new pulmonary rehabilitation program within 60 days of Visit 1. Subjects in the maintenance phase of pulmonary rehabilitation program are not excluded.
14. Treatment with oral, parenteral, or intra-articular corticosteroids within 4 weeks prior to Visit 1.
15. Omalizumab or any other monoclonal or polyclonal antibody therapy taken for any reason within 6 months prior to Visit 1.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2026 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2016-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Ferguson, MD, Principal Investigator — Pulmonary Research Insititute of Southeast Michigan
Locations (174):
- United States (110):
  - Research Site, Andalusia, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Foley, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Flagstaff, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Fresno, California
  - Research Site, Fullerton, California
  - Research Site, Gold River, California
  - Research Site, Lakewood, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Rancho Mirage, California
  - Research Site, San Jose, California
  - Research Site, Westminster, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sebring, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Nampa, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Brownsburg, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Opelousas, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Sunset, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Brockton, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Port Huron, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Plymouth, Minnesota
  - Research Site, Biloxi, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Marlton, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Jackson Heights, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cornelius, North Carolina
  - Research Site, Flat Rock, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Cadiz, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Genoa, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Willoughby, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Scottdale, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Easley, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, Sealy, Texas
  - Research Site, Midvale, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Herndon, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Kingwood, West Virginia
- Argentina (7):
  - Research Site, CABA
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Nueve de Julio
  - Research Site, Ranelagh
  - Research Site, San Miguel de Tucumán
- Bulgaria (10):
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Sandanski
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Velingrad
- Research Site, Santiago, Chile
- Czechia (9):
  - Research Site, Beroun
  - Research Site, Brandýs nad Labem
  - Research Site, Krnov
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Strakonice
  - Research Site, Žatec
- Germany (8):
  - Research Site, Aschaffenburg
  - Research Site, Bad Lippspringe
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Hanover
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Magdeburg
- Mexico (5):
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, San Juan del Río
  - Research Site, Sonora
- Poland (15):
  - Research Site, Aleksandrów Łódzki
  - Research Site, Bialystok
  - Research Site, Bielsk Podlaski
  - Research Site, Bydgoszcz
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Skarżysko-Kamienna
  - Research Site, Turek
  - Research Site, Zabrze
  - Research Site, Żnin
- Research Site, San Juan, Puerto Rico
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eManzimtoti
  - Research Site, Gauteng
- Spain (4):
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Loja (Granada)
  - Research Site, Zaragoza

REFERENCES:
- See also: Symbicort RISE Revised CSP 3 4 FINAL Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2887&filename=Symbicort_RISE_Revised_CSP_3_4_FINAL_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number in the protocol section denotes the number of patients screened into the trial. Out of these 2026 patients screened, 1219 patients were randomized into the trial. This explains the discrepancy in patient number.
Period: Overall Study
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Started | 606 | 613
Completed | 567 | 548
Not Completed | 39 | 65
Not completed — Withdrawal by Subject | 25 | 39
Not completed — Screen failure | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Progressive disease | 0 | 2
Not completed — Other | 5 | 12
Not completed — Lack of Efficacy | 0 | 1
Not completed — Death | 4 | 4
Not completed — Adverse Event | 3 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set including all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler | Total
Number analyzed (Participants) | 606 | 613 | 1219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (8.65) | 63.9 (8.67) | 63.5 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 270 | 521
  Male | 355 | 343 | 698
FEV1 post-bronchodilator categories [Number; unit: Participants]
  <30% | 59 | 54 | 113
  >=30% to <50% | 234 | 247 | 481
  >=50% to <=70% | 307 | 308 | 615
  >70% | 4 | 3 | 7
Number of exacerbations during 2 - 52 weeks prior to enrollment [Number; unit: Participants]
  1 | 430 | 448 | 878
  2 | 136 | 117 | 253
  3 | 29 | 28 | 57
  4 | 7 | 13 | 20
  5 | 2 | 6 | 8
  6 | 0 | 1 | 1
  7 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Moderate and Severe COPD Exacerbations Defined as: Worsening of ≥2 Major Symptoms or Worsening of 1 Major Symptom Together With ≥1 Minor Symptom for ≥2 Consecutive Days
Description: The annual COPD exacerbation rate was analyzed and compared between two arms.
  Annual exacerbation rate for each subject is defined as number of exacerbations divided by duration of randomized treatment period in years.
  The annual COPD exacerbation rate of Symbicort group was compared with annual rate of Formoterol group. The rate ratio of Symbicort vs. Formoteroal was assessed by a negative binomial model.
  Exacerbations, that met the modified Anthonisen criteria and duration ≥2 days were classified as moderate and severe exacerbations.
  Moderate exacerbation: treatment of symptoms with systemic corticosteroids (≥3 days) and/or antibiotics.
  Severe exacerbation: symptoms that require hospitalization (including >24 hours in ED/urgent care setting).
Time Frame: Randomization at Week 0 to End of Treatment (EoT) W 26
Population: Full analysis set including all randomized subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: COPD exacerbations per year
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 606 | 613
COPD exacerbations per year | 0.85 [0.70 to 1.03] | 1.12 [0.93 to 1.35]
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0059, Negative binomial model; Rate ratio = 0.76, 95% CI 2-sided [0.62 to 0.92]

2. Secondary Outcome: Number of Patients With Moderate or Severe COPD Exacerbation.
Description: The number of patients who developed moderate or severe COPD exacerbation during treatment period were reported. Cox proportional hazards regression model was fitted to data to compare the two treatment arms .
  The hazard ratio and 95% CI were estimated.
Time Frame: From randomzation to EoT W 26
Measure: Number; unit: Participants
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 606 | 613
Participants | 171 | 204
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0164, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.64 to 0.96]

3. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ)
Description: SGRQ is a standardized, self-administered tool for measuring impaired health and perceived wellbeing in respiratory diseases; a validated electronic version of the questionnaire in the relevant validated languages was used in this study.
  The questionnaire contains 50 items divided into three dimensions (Symptoms, Activity and Impact).
  Each of the three dimensions of the questionnaire is scored separately in the range from 0 to 100:
  zero (0) score indicating no impairment of quality of life.
  The total SGRQ score ranging from 0 to 100 is a summary score utilizing responses to all items calculated using weights attached to each item of the questionnaire.
  Higher scores indicate poorer health and change of 4 units in the SGRQ has been determined to be the threshold for a clinically relevant change in health status.
  The change from baseline was statistically summarized and compared between two arms in a mixed model.
Time Frame: From Run-in W -4 to EoT W 26
Population: The change from baseline in SGRQ were analyzed on randomized patients with a baseline SGRQ and at least one post-baseline value. Among 1219 patients who were randomized, only 589 patients in Symbicort group and 593 patients in Formoterol group had valid data and included in analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 589 | 593
scores on a scale | -0.855 (8.941) | 0.442 (9.457)
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0070, Mixed Models Analysis; Mean Difference (Final Values) = -1.343, 95% CI 2-sided [-2.318 to -0.368]

4. Secondary Outcome: Pre-dose/Pre-bronchodilator FEV1 at the Study Site
Description: FEV1 from pre-dose spirometry is a measurement of lung function. The change from baseline on pre-dose FEV1 was summarized and compared between Symbicort and Formoterol groups using a mixed model.
Time Frame: From Run-in W -4 to EoT W 26
Population: The change from baseline in pre-dose FEV1 were analyzed on randomized patients with a baseline pre-dose FEV1 and at least one post-baseline value. Among 1219 patients who were randomized, only 588 patients in Symbicort group and 589 patients in Formoterol group had valid data and included in analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 588 | 589
L | 0.008 (0.210) | -0.025 (0.198)
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0091, Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [0.008 to 0.053]

5. Secondary Outcome: Total Rescue Medication Use (Average Puffs/Day)
Description: Use of rescue medication is a measure of symptoms that need to be treated with a short-acting bronchodilator.
  The average daily use across the observation period was used for analysis. Change from baseline was summarized and compared between two arms using a mixed model.
Time Frame: From Run-in W -4 to EoT W 26
Population: The change from baseline on rescue medication use were analyzed on randomized patients with a baseline and a post-baseline value. Among 1219 patients who were randomized, only 602 patients in Symbicort group and 607 patients in Formoterol group had valid data and included in analysis.
Measure: Mean (Standard Deviation); unit: puffs/day
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 602 | 607
puffs/day | 0.135 (1.248) | 0.343 (1.456)
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0082, ANCOVA; Mean Difference (Final Values) = -0.203, 95% CI 2-sided [-0.353 to -0.053]

6. Secondary Outcome: Nights With Awakening Due to COPD
Description: Nighttime awakening due to COPD symptoms correspond to the severity of nocturnal symptoms from COPD.
  The average number of awakening per night over the treatment period was analyzed. It was derived as the number of night with awakening divided by the total number of nights with data in the recording period. Change from baseline period on awakening was summarized and compared between two arms using a mixed model.
Time Frame: From Run-in W -4 to EoT W 26
Population: The change from baseline on awakening were analyzed on randomized patients with a baseline and a post-baseline value. Among 1219 patients who were randomized, only 603 patients in Symbicort group and 610 patients in Formoterol group had valid data and included in analysis.
Measure: Mean (Standard Deviation); unit: awakening/night
Arm/Group | Symbicort pMDI | Formoterol Turbuhaler
Number analyzed (Participants) | 603 | 610
awakening/night | -0.007 (0.173) | 0.021 (0.195)
Statistical Analysis 1: Comparison: Symbicort pMDI vs Formoterol Turbuhaler; Test type: Superiority or Other; p = 0.0048, ANCOVA; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.048 to -0.009]

ADVERSE EVENTS:
Time Frame: During the randomized treatment period, ie from first treatment to one day after the last treatment.
Arm/Group | Formoterol 4.5 ug x2 Bid | Symbicort 160/4.5 ug x2 Bid
Serious Adverse Events (participants affected / at risk) | 63/613 | 49/605
Other Adverse Events (participants affected / at risk) | 56/613 | 38/605
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formoterol 4.5 ug x2 Bid (N=613) | Symbicort 160/4.5 ug x2 Bid (N=605)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (2)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 20 (22)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formoterol 4.5 ug x2 Bid (N=613) | Symbicort 160/4.5 ug x2 Bid (N=605)
Nasopharyngitis (Infections and infestations) | 32 (35) | 30 (34)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No